CLINICAL TRIAL: NCT01726556
Title: A Randomized Controlled Trial of Rigid Versus Semirigid Thoracoscopy in the Evaluation of Exudative Pleural Effusions
Brief Title: A Trial of Rigid Versus Semirigid Thoracoscopy in the Evaluation of Exudative Pleural Effusions
Acronym: RISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Sahajal Dhooria, Senior Resident, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 1Trg-PG-2012/5054
Record Dates: First submitted 2012-11-07; First posted 2012-11-15 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Pleurisy With Effusion
Keywords: Pleural effusion; Semirigid thoracoscopy; Rigid thoracoscopy
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rigid thoracoscopy (Active Comparator): Rigid thoracoscopy would be done using a rigid thoracoscope manufactured by Richard Wolf GmbH, Knittlingen, Germany.
  Interventions: Device: Rigid thoracoscope (Richard Wolf GmbH, Knittlingen, Germany)
- Semirigid thoracoscopy (Active Comparator): The semirigid thoracoscope employed is a model LTF-160Y1, manufactured by Olympus Medical Systems Corporation, Tokyo, Japan.
  Interventions: Device: Semirigid thoracoscope (model LTF-160Y1, Olympus, Japan)

INTERVENTIONS:
Device: Rigid thoracoscope (Richard Wolf GmbH, Knittlingen, Germany) — Pleuroscopy using a rigid thoracoscope manufactured by Richard Wolf GmbH, Knittlingen, Germany
  Arms: Rigid thoracoscopy
Device: Semirigid thoracoscope (model LTF-160Y1, Olympus, Japan) — Pleuroscopy using a semirigid thoracoscope model LTF-160Y1, manufactured by Olympus Medical Systems Corporation, Tokyo, Japan
  Arms: Semirigid thoracoscopy

SUMMARY:
Rigid thoracoscopy is an established procedure for the performance of pleural biopsies for undiagnosed pleural effusions. The semirigid thoracoscope is a relatively new instrument designed for the same purpose which is claimed to be more user-friendly. The two devices have not been compared in a head-to-head trial in published literature. The investigators attempt to conduct a randomised comparative trial between the two devices.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an exudative (as defined by Light's criteria) pleural effusion of unknown etiology after a microbiological (namely gram stain and acid fast bacillus stain) and cytological examination

Exclusion Criteria:

* Significant hypoxemia on room air
* Hemodynamic instability
* Significant cardiac disease (known myocardial infarction in last 6 weeks or presence of unstable angina)
* Refractory cough
* Lack of pleural space due to adhesions
* Uncorrected coagulopathy

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield of thoracoscopic biopsy by intention to treat analysis | 3 months
  The proportion of patients where thoracoscopic pleural biopsy yielded a diagnosis that was consistent with the present clinical picture and the further follow-up of the patients, would be calculated and compared between the two arms

SECONDARY OUTCOMES:
Yield of biopsies successfully completed | 3 months
  The diagnostic yield of only those procedures would be considered separately where a biopsy could be successfully done and compared between the two arms
Complications | 3 months
  Number of major and minor complications encountered in the two arms
Scar size | At the end of the procedure
  Scar size (in mm) in the longest axis
Biopsy size | At the end of the procedure
  Biopsy size (in mm) in the longest axis

OTHER OUTCOMES:
Use of sedation and analgesia during the procedure | At the end of procedure
  The quantity of drugs used for sedation and analgesia during the procedure would be recorded and compared between the two arms
Operators' experience characteristics | At the end of the procedure
  These would include, on a numerical scale of 0 to 100, the operator's grading of the following characteristics: quality of thoracoscopic image, ease of maneuvering, ease of taking a biopsy and the operator's expectation that the biopsy will reveal a definitive histological diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Ritesh Agarwal, MD, DM, Principal Investigator — PGIMER, Chandigarh
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, Chandigarh, India

REFERENCES:
- [Derived] Dhooria S, Singh N, Aggarwal AN, Gupta D, Agarwal R. A randomized trial comparing the diagnostic yield of rigid and semirigid thoracoscopy in undiagnosed pleural effusions. Respir Care. 2014 May;59(5):756-64. doi: 10.4187/respcare.02738. Epub 2013 Oct 8. PMID 24106326